CLINICAL TRIAL: NCT04629079
Title: Lung Cancer Detection Using Blood Exosomes and HRCT- Improving the Early Detection of Lung Cancer by Combining Exosomal Analysis of Hypoxia With Standard of Care Imaging
Brief Title: Improving the Early Detection of Lung Cancer by Combining Exosomal Analysis of Hypoxia With Standard of Care Imaging
Acronym: LungExoDETECT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: King's College London (Other)
Responsible Party: Sponsor
Other Study IDs: 261766
Record Dates: First submitted 2020-10-30; First posted 2020-11-16 (Actual); Last update posted 2020-11-16 (Actual); Status verified 2020-10

CONDITIONS: Lung Cancer
Keywords: Early detection
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples processed for serum, plasma and PBMC extraction
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This project aims to validate exosomal assays that are based on hypoxia detection as potential biomarkers of early detection. The study analysis will determine whether the assay can detect clinical lung cancer at the time of imaging and interval cancers during subsequent follow up. The study aims to establish preliminary sensitivity/specificity data for the "combined CT/exosomal risk stratification marker" and provide initial data on the potential association of the "combined CT/exosomal risk score" with the subsequent cancer progression and treatment response.

DETAILED DESCRIPTION:
Lung cancer is the leading cause of cancer deaths. Screening for early detection of cancer at an early stage reduces cancer deaths and therefore improves prognosis. The National Lung Screening Trial (NLST), for instance, showed that CT screening increases the early detection rate, and reduces mortality. However, drawbacks include over-diagnosis, false-positive results, psychological distress and cost. Therefore, lung cancer screening is not recommended or available within the NHS.

Diagnosis of lung cancer is currently based on a combination of scans and tissue biopsy. The invasive nature of current diagnostic procedures limits their application. To improve the efficacy and cost effectiveness of screening in early detection of lung cancer, additional, complementary and non-invasive methods, such as circulating biomarkers, should be evaluated. Our novel exosomal assay (taken from a blood sample) when combined with CT, may improve the current accuracy of lung cancer detection, especially that of a worse clinical prognosis. Improvement in the accuracy of detection and/or prediction of future disease by performing the combined imaging exosome test will cause a paradigm shift. Moving towards the identification of blood tests can help increase confidence about follow-up decisions and shorten the interval before biopsy.

This prospective cohort study will recruit patients referred to secondary care for the investigation of clinical symptoms or signs suspicious of lung cancer.

The study will run between 2020 and 2024 (two-year active recruitment and two-year follow up).

Participants will have a single assay of blood taken on one occasion in the lung clinic by trained staff.

Participants will have normal standard of care chest CT scans and this data will be used.

All participants will be actively followed for 3 months and then those with nodules, revealed by CT Scan, at 3 monthly intervals. Longitudinal clinical data will be collected on the investigations, diagnoses and outcomes of all study patients.

Data will be collected on date, type and results of imaging and biopsy investigations including nodule size and progression.

For those diagnosed with lung cancer, data on tumour size, stage, type and other markers) will be recorded together with treatment response and date of death, where this occurs within the study.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age
* Suspected clinical diagnosis of lung cancer
* Able to provide informed consent

Exclusion Criteria:

-Synchronous other cancer types.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will include patients who have been referred to the Lung Cancer Clinic and Multi- Disciplinary Team (MDT) at The Lister, Hertford County and New QEII Hospitals for investigation of suspected lung cancer.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2020-10-23 (Actual); Primary Completion 2022-10-23 (Estimated); Study Completion 2024-10-23 (Estimated)

PRIMARY OUTCOMES:
Describe the range of exosomal expression of P4HA1 in participants being clinically assessed for a suspected lung cancer diagnosis and compare the range of expression between the cancer and non-cancer participant population. | Through study completion, an average of 2 years.
  Describe the expression of hypoxia- response element (HRE) responsible protein P4HA1 utilising a hypoxia-reporting cancer exosomal assay in participants being clinically assessed for suspected lung cancer.

SECONDARY OUTCOMES:
Describe the range of expression of precursor microRNA in exosomes derived from participants being clinically assessed for suspected lung cancer and compare the range of expression between the cancer and non-cancer participant population. | Through study completion, an average of 2 years.
  Utilise exosome-based assessment of pre-microRNA processing to inform the development of a hypoxia gene signature for the early detection of lung cancer.
Develop a combined risk score combining multi-dimensional parameters to discriminate between cancer cases and non-cancer cases. | Through study completion, an average of 2 years.
  To develop a combined risk prediction model to support the early diagnosis of lung cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Thida Win, MD, Principal Investigator — Lister Hospital
Locations (1):
- Borthwick Research Unit, Lister Hospital, Stevenage, United Kingdom

IPD SHARING:
Plan to Share IPD: No